CLINICAL TRIAL: NCT00690248
Title: Prevalence of Depressive Symptoms in Manic Episodes of Bipolar Patients: an Observational Study
Brief Title: Depressive Symptoms in Acute Manic Episode
Acronym: MM1
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Teresa Díez, PhD, Local MC Neuroscience Therapeutic Area Manager, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NES-DUM-2007/5
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Bipolar Disorder
Keywords: Acute mania; Bipolar disorder; depressive symptoms; mixed mania
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Bipolar patients admitted to a psychiatric Unit due to an acute mania episode.

SUMMARY:
Observational, non-interventional, transversal, multicenter, open label (No treatment is involved). The primary objective is to detect the prevalence of depressive symptoms in bipolar patients admitted to a psychiatric Unit due to an acute mania episode. Secondary objectives include 1) to evaluate, the relationship between depressive symptoms and severity of mania; 2) to evaluate, the relationship between depressive symptoms and anxiety; 3) to evaluate, the relationship between depressive symptoms and psychotic symptoms; 4) to evaluate, the relationship between depressive symptoms and insight; 5) to evaluate, the relationship between depressive symptoms and clinical global impression; 6) to evaluate, the relationship between depressive symptoms and previous treatment with antipsychotics (whatever the antipsychotic was); 7) to evaluate, the relationship between depressive symptoms and length of admission; 8) to evaluate factors (demographic, evolution…) which could be involved in the presence of depressive symptoms within an acute manic episode; 9) to evaluate, the difference on the initial prescription due to the detection of depressive symptoms; 10) to evaluate, if exists, differences on the previous psychiatric diagnosis in patients with and without depressive symptoms. The primary endpoint is score of the MADRS (Montgomery-Asberg Depression Rating Scale) in bipolar patients with acute mania

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of Bipolar Disorder based on DSM-IV-TR
* Patients admitted to an acute inpatient psychiatric Unit due to an acute manic episode (as defined in DSM-IV_TR)
* Provision of written informed consent.
* Total score in Young Mania Rating Scale >=20
* Able to understand and comply with the requirements of the study

Exclusion Criteria:

* Mental retardation
* Patients with manic symptoms are due to substance use, based in the investigator opinion
* Patients with unstable organic diseases, who are not receiving adequate treatment, according the investigator opinion.
* Participation in a trial with drugs within 4 weeks of enrolment into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: bipolar patients admitted to a psychiatric Unit due to an acute mania episode.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Score of the MADRS (Montgomery-Asberg Depression Rating Scale) in bipolar patients with acute mania. | once during study

SECONDARY OUTCOMES:
Mania symptoms measured with YMRS (Young Mania Rating Scale). | once during study
Anxiety symptoms measures with HARS (Hamilton Anxiety Rating Scale). | once during study
Psychotic symptoms measured with BPRS (Brief Psychosis Rating Scale). | once during study
Clinical status and improvement measured with CGI-BP (Clinical Global Impression - Bipolar scale). | once during study
Days of hospitalization, MADRS (6 items) | once during study
Hamilton Depression Rating Scale (5 items) | once during study
Scale of Unawareness of Mental Disorders (SUMD) | once during study

CONTACTS AND LOCATIONS:
Locations (34):
- Spain (34):
  - Research Site, A Coruña
  - Research Site, Alcoy
  - Research Site, Algeciras
  - Research Site, Almería
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Córdoba
  - Research Site, Granada
  - Research Site, Las Palmas
  - Research Site, Logroño
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Osuna
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Plasencia
  - Research Site, Ponferrada
  - Research Site, Pontevedra
  - Research Site, Salamanca
  - Research Site, San Juan (Alicante)
  - Research Site, Sant Boi de Llobregat
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Santander
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Teruel
  - Research Site, Toledo
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Vitoria-Gasteiz
  - Research Site, Zamora
  - Research Site, Zaragoza